CLINICAL TRIAL: NCT03395353
Title: A Long-term Safety Study of Duloxetine Hydrochloride in the Treatment of Japanese Children and Adolescents With Depressive Disorder
Brief Title: A Study of Duloxetine (LY248686) in the Treatment of Japanese Children and Adolescents With Depressive Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Shionogi (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16916; F1J-JE-HMHF (Other: Eli Lilly and Company); 1702A3632 (Other: Shionogi)
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Duloxetine hydrochloride (Experimental): Duloxetine hydrochloride administered orally.
  Interventions: Drug: Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine Hydrochloride — Administered orally
  Other Names: LY248686

SUMMARY:
The purpose of this long-term study is to evaluate the safety and efficacy of duloxetine hydrochloride in Japanese children and adolescents with depressive disorder.

ELIGIBILITY:
* a) Participants extended from B058(1701A3631) study.
* b) New participants.

Inclusion Criteria

* a) Participants who have completed 7 weeks of dosing in the B058(1701A3631) study and give signed informed consent to continue duloxetine administration in this study.
* b) Participants diagnosed with Major Depressive Disorder or persistent depressive disorder and completely meet the criteria of major depressive episode as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) with the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) ver.7.0.2.
* b) Participants whose incipient age of depression was ≥7 years old.

Exclusion Criteria:

* a, b) Have a current or previous diagnosis (DSM-5) of the following as judged by the investigator:

  * Neurodevelopmental disorders
  * Schizophrenia spectrum and other psychotic disorders
  * Bipolar and related disorders
  * Trauma and stressor-related disorders
  * Disruptive · Impulse Control · and Conduct disorders
* a, b) Have a current diagnosis (DSM-5) of the following as judged by the investigator:

  * Obsessive-compulsive and related disorders
  * Anorexia nervosa, Bulimia nervosa, Binge-eating disorder
  * Sleep-wake disorders
  * Neurocognitive disorders
  * Disruptive mood dysregulation disorder
* a, b) Have personality disorders, in the judgment of the investigator.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2020-07-04 (Actual); Study Completion 2020-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (1):
- Shionogi, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shibata RY, Kubota R, Uenaka K, Kaibara A, Wajima T. Population pharmacokinetics of duloxetine in Japanese pediatric patients with major depressive disorder. Drug Metab Pharmacokinet. 2023 Aug;51:100496. doi: 10.1016/j.dmpk.2023.100496. Epub 2023 Feb 15. PMID 37244205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 59 and 64 subjects, respectively, were enrolled consecutively from the placebo- and duloxetine-group in the preceding study 1701A3631/F1J-JE-B058, NCT03315793. 28 new participants were also enrolled.
Groups:
- Duloxetine: 20 mg Duloxetine was administered every day for 1 week. Then 40 mg Duloxetine was administered for 1 week. Then flexible doses of 40 mg or 60 mg Duloxetine were administered for 48 weeks till end of treatment period. Lower doses of Duloxetine were administered for 1 to 2 weeks during tapering off period.
Period: Overall Study
Arm/Group | Duloxetine
Started | 151
Received At Least 1 Dose of Study Drug | 150
Completed | 64
Not Completed | 87
Not completed — Adverse Event | 20
Not completed — Protocol Violation | 1
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 24
Not completed — Discontinued visit | 1
Not completed — Refrain from visit due to COVID-19 | 1
Not completed — Physician Decision | 4
Not completed — Early termination of overall study | 33

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug. One participant received no dose of study drug and was not included in the analysis.
Arm/Group | Duloxetine
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 150
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 150
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 150

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs), Drug Related Adverse Events (ADRs) or Any Serious Adverse Events (SAEs)
Description: A summary of AEs, ADRs (considered by the investigator) and SAEs is located in the Reported Adverse Events module. An AE was included if the onset date is on or after the first dose of study drug and within 7 days after the last dose, or it is consecutive from the preceding study at the initiation of study drug administration in this study.
Time Frame: Baseline through Week 53
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 150
percentage of participants
  Serious Adverse Event | 2
  Adverse Event including Serious Adverse Event | 89.3
  Drug-Related Adverse Event | 73.3

2. Secondary Outcome: Change From Baseline on the Children's Depression Rating Scale-Revised (CDRS-R)
Description: Children's Depression Rating Scale-Revised (CDRS-R) Total score measures the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning and higher numbers indicate a higher degree of depression. The total sum of scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, scores of 40 to 60 indicate moderate depression, and scores greater than 60 indicate severe depression.
Time Frame: Baseline, Week 50
Population: All enrolled participants who received at least one dose of study drug and had at least 1 post-dose CDRS-R Total score. Missing values due to discontinuation of study or missing data were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 150
units on a scale | -12.8 (16.7)

3. Secondary Outcome: Change From Baseline on the Clinical Global Impression-Severity of Illness (CGI-S)
Description: CGI-S measures severity of illness at the time of assessment compared with start of treatment with scores ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Baseline, Week 50
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 150
units on a scale | -0.9 (1.3)

4. Secondary Outcome: Pharmacokinetics (PK): Trough Concentration of Duloxetine
Description: Trough concentrations of duloxetine are defined as the plasma concentrations in 18 - 30 hours post the previous dose. PK samples were obtained from each subject from Week 4 to the end of treatment period (Week 50) for analysis of steady state duloxetine concentrations. If duloxetine dose changed, PK samples were taken after 2 week or more administration of the new dose. Principally 1 or 2 blood samples were drawn from each subject at pre-dose for trough concentrations.
Time Frame: Week 4 through Week 50
Population: All enrolled participants who received at least 1 dose of study drug. 512 plasma concentrations were from 141 subjects, 20 of which were excluded due to discontinuation, overdose and subjects being non-Japanese. 492 concentration values from 136 Japanese subjects were included in the analysis. Of the 492 concentration values, 133 from 106 subjects were trough concentrations. Sum of subjects(3, 47, 6, 54) is 110, 4 more than 106, as 4 subjects of 12-17 years old are redundant in 40mg and 60mg.
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: Trough Concentration
Groups:
- Duloxetine 40 mg (9 to 11 Years Old): Trough concentrations of duloxetine 40mg were obtained from 9 to 11 year olds. Trough concentrations are defined as the plasma concentrations 18 to 30 hours after the last administration of duloxetine.
- Duloxetine 40 mg (12 to 17 Years Old): Trough concentrations of duloxetine 40mg were obtained from 12 to 17 year olds. Trough concentrations are defined as the plasma concentrations 18 to 30 hours after the last administration of duloxetine.
- Duloxetine 60 mg (9 to 11 Years Old): Trough concentrations of duloxetine 60mg were obtained from 9 to 11 year olds. Trough concentrations are defined as the plasma concentrations 18 to 30 hours after the last administration of duloxetine.
- Duloxetine 60 mg (12 to 17 Years Old): Trough concentrations of duloxetine 60mg were obtained from 12 to 17 year olds. Trough concentrations are defined as the plasma concentrations 18 to 30 hours after the last administration of duloxetine.
Arm/Group | Duloxetine 40 mg (9 to 11 Years Old) | Duloxetine 40 mg (12 to 17 Years Old) | Duloxetine 60 mg (9 to 11 Years Old) | Duloxetine 60 mg (12 to 17 Years Old)
Number analyzed (Participants) | 3 | 47 | 6 | 54
Number analyzed (Trough Concentration) | 4 | 52 | 7 | 70
ng/mL | 8.51 (7.22) | 18 (15.2) | 33.4 (30.7) | 39.5 (52.1)

ADVERSE EVENTS:
Time Frame: Baseline to 53 Weeks
Description: All participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Duloxetine
All-Cause Mortality (participants affected / at risk) | 0/150
Serious Adverse Events (participants affected / at risk) | 3/150
Other Adverse Events (participants affected / at risk) | 134/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=150)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=150)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Hyperacusis (Ear and labyrinth disorders) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 1 (1)
Blepharitis allergic (Eye disorders) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Myopia (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 46 (56)
Constipation (Gastrointestinal disorders) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Dental caries (Gastrointestinal disorders) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 7 (8)
Stomatitis (Gastrointestinal disorders) | 7 (9)
Vomiting (Gastrointestinal disorders) | 6 (8)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Oral pruritus (Gastrointestinal disorders) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1)
Malaise (General disorders) | 8 (8)
Withdrawal syndrome (General disorders) | 5 (5)
Thirst (General disorders) | 4 (4)
Feeling abnormal (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 4 (4)
Anovulatory cycle (Endocrine disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 50 (64)
Gastroenteritis (Infections and infestations) | 5 (5)
Influenza (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Dermatitis infected (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Skin bacterial infection (Infections and infestations) | 1 (1)
Malassezia infection (Infections and infestations) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1)
Purulence (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3)
Wound (Injury, poisoning and procedural complications) | 2 (2)
Chilblains (Injury, poisoning and procedural complications) | 1 (2)
Ear canal abrasion (Injury, poisoning and procedural complications) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 1 (1)
Weight increased (Investigations) | 4 (4)
Blood bilirubin increased (Investigations) | 3 (4)
Blood pressure increased (Investigations) | 3 (3)
Heart rate increased (Investigations) | 3 (4)
Weight decreased (Investigations) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 2 (2)
Blood uric acid increased (Investigations) | 2 (2)
Liver function test increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (2)
Haemoglobin decreased (Investigations) | 1 (1)
Protein total decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Protein urine present (Investigations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Somnolence (Nervous system disorders) | 42 (48)
Headache (Nervous system disorders) | 20 (25)
Dizziness (Nervous system disorders) | 17 (18)
Dizziness postural (Nervous system disorders) | 5 (5)
Paraesthesia (Nervous system disorders) | 2 (2)
Akathisia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Irregular sleep wake rhythm disorder (Nervous system disorders) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 18 (23)
Insomnia (Psychiatric disorders) | 3 (3)
Sleep disorder (Psychiatric disorders) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 3 (3)
Irritability (Psychiatric disorders) | 2 (2)
Suicide attempt (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Hallucinations, mixed (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Middle insomnia (Psychiatric disorders) | 1 (1)
Neurosis (Psychiatric disorders) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Trichotillomania (Psychiatric disorders) | 1 (1)
Affect lability (Psychiatric disorders) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3)
Menstruation irregular (Reproductive system and breast disorders) | 2 (2)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1)
Premenstrual syndrome (Reproductive system and breast disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Colour blindness (Congenital, familial and genetic disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 6 (7)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT03395353/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT03395353/SAP_001.pdf